CLINICAL TRIAL: NCT01855217
Title: Pilot Study on the Pharmacodynamics of Sugammadex in Morbidly Obese Patients: Reversal of Deep Neuromuscular Blockade
Acronym: MOS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, A. Houwink, MD, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: NL40732.100.12
Record Dates: First submitted 2013-04-02; First posted 2013-05-16 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Neuromuscular Blockade
Keywords: morbid; obesity; sugammadex; pharmacodynamics
MeSH Terms: conditions — Obesity | interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sugammadex total body weight (Active Comparator): 1 mg/kg total body weight
  Interventions: Drug: Sugammadex
- Sugammadex ideal body weight (Active Comparator): 1 mg /kg ideal body weight
  Interventions: Drug: Sugammadex
- placebo (Placebo Comparator): placebo 0,9% NaCl
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sugammadex — 1 mg/kg total BW based sugammadex reversal of deep block
  Other Names: Bridion
  Arms: Sugammadex total body weight
Drug: Sugammadex — 1 mg/kg ideal BW based sugammadex reversal of deep block
  Other Names: Bridion
  Arms: Sugammadex ideal body weight
Drug: Placebo — 0,9% NaCl
  Other Names: 0,9% NaCl
  Arms: placebo

SUMMARY:
Should the dose of sugammadex in morbid obese patients be calculated on the real body weight or the ideal body weight?

To study the pharmacodynamics of sugammadex in morbidly obese patients by comparing 1 mg/kg IBW versus 1 mg/kg TBW versus placebo.

DETAILED DESCRIPTION:
Background of the study:

Morbidly obese patients selected for elective bariatric surgery have major anesthetic concerns. The risks include a difficult airway, difficult mask ventilation, hypoxemia, pre-existent restrictive and obstructive lung disease and residual anesthetics postoperatively due to their body habitus. In this research the investigators will focus on reversal of neuromuscular blockade to give the patient full muscle strength. Sugammadex is a A-cyclodextrin designed to encapsulate rocuronium bromide, a frequently used non-depolarizing neuromuscular blocking agent. Sugammadex provides rapid reversal of neuromuscular blockade by this encapsulation. Based on the available literature, it can be concluded that limited information is available on the use of sugammadex in morbidly obese patients. While the degree of obesity varies within the available studies, in general, the studied patients are less obese compared to the population that is currently undergoing bariatric surgery. The pharmaceutical company that produces sugammadex states that it should be dosed based on the total body weight (TBW) in all adults, regardless of the presence of obesity. However, rocuronium bromide in morbidly obese patients is dosed on ideal body weight (IBW). Therefore, the investigators hypothesize that sugammadex can be dosed based on ideal body weight instead of total body weight in morbidly obese patients. This is also relevant in economic perspective since the costs of sugammadex are high.

Objective of the study:

To study the pharmacodynamics of sugammadex in morbidly obese patients by comparing 1 mg/kg IBW versus 1 mg/kg TBW versus placebo

Study design:

This is a double-blind randomized, placebo controlled study which will be performed in morbidly obese patients with a BMI > 40 kg/m2 undergoing bariatric surgery . Patients about to undergo bariatric surgery will be approached and asked to participate. Before induction of anesthesia, a neuromuscular train-of-four (NMT)(type M-NMT-00=00, Datex Engstrom) will be applied over the ulnar nerve by use of surface electrodes. By placing two electrodes over the nervus ulnaris and giving four pulses of 0,2 ms duration delivered at a frequency of 2 Hz every 15 seconds it will give a muscle twitch. With the Train-of-four (TOF) the investigators can measure the neuromuscular response of the adductor pollicis muscle and calculate the neuromuscular blockade over time ( TOF percentage). The TOF percentage will be measured from induction of anesthesia until the end of surgery. According to a standardized anesthesia protocol, propofol (2.5 mg kg-1) and fentanyl 250microgram will be given for induction of anesthesia, upon which the NMT will be calibrated and the resultant force of contraction of the adductor pollicis muscle is recorded. This is followed by rocuronium 0,6 mg/kg based on IBW and after the TOF ratio has come 0%, tracheal intubation will take place and mechanical ventilation will be initiated by the attending anesthesiologist. Patients then receive either sugammadex 1 mg/kg based on ideal body weight (IBW) or 1mg/kg based on total body weight (TBW) or placebo 0,9% NaCl as a bolus injection in a double blind fashion. During surgery, the attending blinded anesthesiologist is allowed to give additional bolus of 10 mg atracurium whenever the neuromuscular block is inadequate in his opinion or the TOF ratio exceeds 50%. Atracurium is not a aminosteroidal neuromuscular blocking agent and can still be used in patients within unlimited hours after use of sugammadex, as it will not be encapsulated by sugammadex. Until two hours after the sugammadex dose the patient will be observed in a usual manner in the PACU.

Study population:

25 morbidly obese patients with a Body Mass Index > 40 kg/m2 who are undergoing bariatric surgery will be included (laparoscopic gastric banding, or -bypass surgery or sleeve-gastrectomy) Inclusion criteria: - Body Mass Index > 40 kg/m2 - 18-65 years old - American Society of Anaesthesiologists (ASA) physical status II to III Exclusion criteria: - Renal insufficiency identified by GFR < 60 ml/min/1.73m2 - Use of sevoflurane since this can enhance neuromuscular blockade - Previous succinylcholine use in the last 24 hours - Use of other medication that can enhance neuromuscular blockade such as aminoglycoside- and polypeptide-antibiotics, lincosamide, acylamino-penicilline-antibiotics, tetracycline, high dose of metronidazol, M.A.O.-inhibitors, kinidine, magnesium, calcium channel blockers, lithium. - Use of other medication that can decrease the neuromuscular blockade such as neostigmine, pyridostigmine, aminopyridinederivates, chronic use of corticosteroids, phenytoïne or carbamazepine, noradrenaline, azathioprine, theofylline, calciumchloride, kaliumchloride. - hypersensitivity (allergic) to sugammadex or any of the preservatives. - Known ejection fraction of less than 35% - Liver failure ( > 3 times the upper limit of normal values) - Pregnancy or breastfeeding

Intervention:

After intubation of the patient either sugammadex or placebo will be given in a double blind fashion. Placebo or sugammadex 1 mg/kg based on IBW or 1 mg/kg based on TBW will be given and the TOF will be measured every 15 second until a ratio of 50% is achieved.

Primary study parameters/outcome of the study:

• Time to TOF 50%

Secondary study parameters/outcome of the study:

• Time to TOF 5% and 25% • Time course of TOF • Relation between TOF% and covariates (TBW, IBW, age, gender etc) • Quality of surgical conditions from muscle relaxation point of view.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: ugammadex is a drug that has been approved to be used in Europe since 2008. Safety data indicates that sugammadex was well tolerated up to the licensed dose of 16 mg/kg. The investigators will give 1 mg/kg based on ideal or total body weight. The use of sugammadex after induction of anesthesia in this dose may lead to insufficient neuromuscular blockade; by using sugammadex, either 1 mg/kg based on IBW or TBW the neuromuscular blockade will be shortened between 7-22 minutes or 5-15 minutes respectively. For the placebo group it is shown that 0,6 mg/kg rocuronium based on ideal body weight will give neuromuscular blockade until a TOF of 50% for 20-40 minutes. As the TOF is continuously measured, the attending anaesthesiologist will monitor neuromuscular blockade using TOF and/or other standard criteria and can consider at any time to administer atracurium to increase neuromuscular blockade during surgery. The perioperative use of the TOF monitor can be considered standard practice

ELIGIBILITY:
Inclusion Criteria:

* must have a Body Mass Index > 40 kg/m2
* must be between 18-65 years old
* must have an American Society of Anesthesiologists (ASA) physical status II to III

Exclusion Criteria:

* Must not have Renal insufficiency identified by GFR < 60 ml/min/1.73m2
* Sevoflurane must not be used since this can enhance neuromuscular blockade
* No previous succinylcholine must be used in the last 24 hours
* No use of other medication that can enhance neuromuscular blockade such as aminoglycoside- and polypeptide-antibiotics, lincosamide, acylamino-penicillin-antibiotics, tetracycline, high dose of metronidazol, M.A.O.-inhibitors, kinidine, magnesium, calcium channel blockers, lithium.
* No use of other medication that can decrease the neuromuscular blockade such as neostigmine, edrofonium, pyridostigmine, aminopyridine derivates, chronic use of corticosteroids, phenytoïne or carbamazepine, noradrenaline, azathioprine, theophylline, calcium chloride, kaliumchloride.
* hypersensitivity (allergic) to sugammadex or any of the preservatives.
* an ejection fraction of less than 35%
* Liver failure
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
50% TOF-recovery after sugammadex | 0-30 minutes
  • Time to Train-of-four 50%

SECONDARY OUTCOMES:
Time to TOF 5% and 25% | 0-30 minutes
  Time course of Train-of-four

OTHER OUTCOMES:
Relation between TOF% and covariates (TBW, IBW, age, gender etc) | 0-30 minutes
  The relation between TOF and covariates will be assessed by using the data on weight, age , gender. As this is a pilot study we can not draw conclusions.
Quality of surgical conditions from muscle relaxation point of view. | 0-end of surgery ( approx 60-90 min)
  The surgeon will be asked to give a score of 1-5 to verify the surgical conditions in a muscle relaxation point of view

CONTACTS AND LOCATIONS:
Overall Officials: H PA van Dongen, Study Director — St. Antonius Hospital
Locations (1):
- Sint Antonius Ziekenhuis, Nieuwegein, Netherlands